CLINICAL TRIAL: NCT00688038
Title: A Study to Determine Correlation of MR Thermal Imaging to Actual Size of Ablation During Laser Therapy of Metastases to Bone
Brief Title: Correlation of MR Thermal Imaging to Actual Size of Ablation During Laser Ablation Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: BioTex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0393; NCI-2011-00518 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Advanced Cancer; Bone Metastases
Keywords: Advanced Cancer; Bone Metastases; Laser Ablation; Magnetic Resonance Thermal Imaging; Laser Induced Thermal Therapy; MRTI; LITT
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser Ablation + MRTI (Experimental): Magnetic resonance thermal imaging = MRTI
  Interventions: Procedure: Laser Ablation; Procedure: Magnetic Resonance Thermal Imaging

INTERVENTIONS:
Procedure: Laser Ablation — Laser ablation procedure taking about 1-3 hours, depending on the size and location of the tumor.
Procedure: Magnetic Resonance Thermal Imaging — MRTI will be used to monitor the temperature within the ablation zone during the laser ablation.
  Other Names: MRTI

SUMMARY:
The goal of this clinical research study is to learn how well magnetic resonance thermal imaging (MRTI) can check the amount of tumor being destroyed using a therapy called laser ablation (a procedure that uses lasers to create heat that is designed to destroy cancer cells).

DETAILED DESCRIPTION:
Laser ablation is designed to destroy tumor tissue with the use of fiber optics that are placed directly into the tumor to deliver laser light energy into the tissue.

In this study, tumor destruction will be checked using MRTI. MRTI is very similar to other MRI techniques, but instead of providing imaging data, MRTI will provide temperature data for cancerous areas in the body during the laser ablation process. If tumor temperature can be measured more accurately, the laser ablation process may be safer.

Laser Ablation and the MRTI Scan:

If you are found to be eligible to take part in this study, on the day you have laser ablation, you will have an intravenous (IV) line placed. You will receive sedation or general anaesthesia (drugs to make you sleep) through a needle in your vein over 1-3 hours to lessen any pain you may have during the procedure. This process will be explained to you.

After receiving the anaesthesia, the following tests and procedures will be performed:

* You will have a limited MRI.
* Your skin will be cleaned and covered with sterile towels and sheets to lower the chance of an infection.
* The doctor will use MRI scans to place a special needle (applicator) into the tumor. This applicator will be used to create heat at a high enough temperature that cells can be destroyed. Small masses may be destroyed in 1 treatment, but larger masses may require that the needle is placed several times. Each heating cycle takes less than 10 minutes.
* During laser ablation, MRTI will be used to monitor the temperature within the ablation zone. The MRTI process is very similar to regular MRI.
* Your heart rate and blood pressure will be measured during the entire procedure.
* The entire procedure may take about 1-3 hours, depending on the size and location of your tumor.

After the procedure is completed, you will be kept in the hospital for 4-6 hours for observation. You will be checked for recovery from the sedation that you received during the procedure. Once you have recovered from the procedure, you will be allowed to leave the hospital. If you have side effects from the procedure, the doctor may decide to keep you in the hospital for a longer time period for observation.

Follow-Up Visits:

After you have completed the procedure, you will return to M. D. Anderson for follow-up visits. About one (1) week after the laser ablation, you will have a physical exam and an X-ray. About one (1) month after the laser ablation, you will have a physical exam and a limited MRI to check the status of the disease.

Length of Study:

You will be considered off-study after the 1-month follow up visit.

This is an investigational study. The laser ablation procedure is an FDA-approved procedure. The devices are commercially available and can be used outside research studies. The investigational part of this study involves using MRTI to check the effect of ablation on the tumor. Up to 24 participants will be enrolled in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with tumor metastases to the skeleton who are referred to interventional radiology for percutaneous ablation
2. Surgery is not a viable or desirable alternative therapy at the time of enrollment
3. Radiation therapy has failed or not indicated or can be safely postponed
4. Symptomatic or asymptomatic tumor size less than or equal to 3 cm in its largest diameter.
5. Performance status is Eastern Cooperative Oncology Group 2 or better in adults
6. Patient is able to undergo MRI
7. Patients at least 18 years of age

Exclusion Criteria:

1. Patients with uncorrectable coagulopathy
2. Patients with pacemaker or defibrillator
3. Patients with metallic prosthesis at the site of the intended ablation
4. Patients with spinal cord compression or epidural tumor extension
5. Patients with vertebral body metastases exhibiting posterior wall destruction
6. Patients with any soft tissue extension of a vertebral tumor
7. Patients with any metastasis that is extrinsically located in vertebra or any long bones of the extremities compromising the cortex
8. Patients with tumors having direct extension or involvement of a joint capsule or a major nerve
9. Patients with Neutropenia (ANC less then 1000) or known active infection
10. Patients unable to undergo conscious sedation
11. Children under 18 years of age will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-05-13 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Correlation of Maximal Dimensions of 60-degree Celsius Isotherm + Ablation Zone Dimensions as determined by MRI | 2 Years
  Magnetic resonance thermal imaging (MRTI) data to determine the correlation between observed temperatures determined from MRTI and the actual size of ablation as determined by post-ablation contrast-enhanced magnetic resonance imaging (MRI) during Laser Induced Thermal Therapy (LITT) of soft tissue metastases in bone.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Ahrar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org